CLINICAL TRIAL: NCT00639990
Title: Effects of PEEP in Brain Injury Patients
Brief Title: Respiratory Mechanics in Brain Injured Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Università degli Studi dell'Insubria (Other)
Responsible Party: Pelosi Paolo, University of Insubria Varese, Italy
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 003; No financial support
Record Dates: First submitted 2008-03-12; First posted 2008-03-20 (Estimated); Last update posted 2008-03-20 (Estimated); Status verified 2008-03

CONDITIONS: Brain Injury; Acute Lung Injury
Keywords: Intraabdominal pressure
MeSH Terms: conditions — Brain Injuries; Acute Lung Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control (Active Comparator): Patients without lung injury and brain injury
  Interventions: Other: PEEP
- Brain No ALI 1 (Experimental): Patients with brain injury and no lung injury within 72 hours from ICU entry
  Interventions: Other: PEEP
- Brain No ALI 2 (Experimental): Patients with brain injury and no ALI after 72 hours from ICU entry
  Interventions: Other: PEEP
- Brain ALI (Experimental): Patients with brain injury and Acute Lung Injury (ALI)
  Interventions: Other: PEEP

INTERVENTIONS:
Other: PEEP — Application of positive end expiratory pressure
  Other Names: No brain injury No ALI
  Arms: Control
Other: PEEP — Application of positive end-expiratory pressure
  Other Names: Brain No ALI 72hrs
  Arms: Brain No ALI 1
Other: PEEP — Application of positive end-expiratory pressure
  Other Names: Brain NO ALI more 72 hrs
  Arms: Brain No ALI 2
Other: PEEP — Application of positive end-expiratory pressure
  Other Names: Brain and ALI
  Arms: Brain ALI

SUMMARY:
The hypothesis is that brain injury patients have alterations of the respiratory system related to intraabdominal pressure. Furthermore application of moderate levels of PEEP may improve respiratory function in these patients.

DETAILED DESCRIPTION:
We investigate the mechanical properties of the respiratory system, partitioned into its lung and chest wall components, the functional residual capacity, the gas-exchange and alveolar recruitment in brain injured patients.

The measurements will be performed under sedation at different levels of PEEP. The following groups will be included: a) control patients withot lung injury and brain injury; b) brain injured patients without lung injury within the first 72 hours; c) brain injured patients without lung injury after 72 hours; d) brain injured patients with lung injury. Brain injury was defined as primary or secondary. Respiratory functional data will be related to intra-abdominal pressure.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female
* Age > 18 yrs
* Mechanical ventilation
* No smoker
* No lung injury at entry
* Brain injury (traumatic or postoperative or spontaneous bleeding) in brain injury group

Exclusion Criteria:

* Pregnancy
* Hemodynamic instability
* Immunodepression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-06; Primary Completion 2008-12 (Estimated); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Improvement of respiratory function with PEEP | 30 min

SECONDARY OUTCOMES:
Relations of respiratory mechanics (lung and chest wall) with intraabdominal pressure | 30 min

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Pelosi, MD, Principal Investigator — University of Insubria, Varese
Locations (1):
- Ospedale di Circolo e Fondazione Macchi, Varese, Varese, Italy